CLINICAL TRIAL: NCT03190772
Title: The Role of Expectations in the Pharmacological Treatment of Depression - An Experimental Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Winfried Rief, Professor Dr., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2017-12k
Record Dates: First submitted 2017-06-14; First posted 2017-06-19 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Major Depressive Episode

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positive placebo group (Experimental): Participants receive a placebo nasal spray. However, they are told that it protects from experiencing negative emotions. Participants watch a film sequence that is supposed to induce sadness.
  Interventions: Other: Placebo nasal spray; Other: Film sequence
- Placebo control group (Placebo Comparator): Participants receive a placebo nasal spray and are told that it is a placebo. Participants watch a film sequence that is supposed to induce sadness.
  Interventions: Other: Placebo nasal spray; Other: Film sequence
- No-treatment control group (Other): Participants do not receive the nasal spray. Participants watch a film sequence that is supposed to induce sadness.
  Interventions: Other: Film sequence

INTERVENTIONS:
Other: Placebo nasal spray — The placebo nasal spray consists of sesame oil and does not contain any active drug.
  Arms: Placebo control group; Positive placebo group
Other: Film sequence — All groups watch the film sequence that is supposed to induce sadness.

SUMMARY:
The study aimes at identifying whether positive expectations have an impact on the way depressive participants experience emotions in the form of sadness.

ELIGIBILITY:
Inclusion Criteria:

* major depression (mild to moderate)
* fluent in German language

Exclusion Criteria:

* bipolar disorder, psychotic disorder, substance dependence
* cardiovascular disease, severe kidney or liver disease, epilepsy
* change of psychotropic medication intake within the last four weeks
* allergic to capsaicin
* allergic to sesame oil
* students in medicine, pharmacy, or psychology in their third year or older
* completed studies in medicine, pharmacy or psychology

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Sadness | Directly after watching the film sequence, no follow-up assessments
  Items of PANAS-X

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Professor, Principal Investigator — Philipps University Marburg
Locations (2):
- Germany (2):
  - Justus Liebig University Gießen, Giessen, Hesse
  - Philipps University Marburg, Marburg, Hesse

IPD SHARING:
Plan to Share IPD: No